CLINICAL TRIAL: NCT00762723
Title: A Comparison of Clinical Outcomes Comparing Fixed-angle, Variable-angle, and Hybrid Screw Configuration for the Trinica(R) Anterior Lumbar Plate System
Brief Title: Clinical Outcomes of the Trinica(R) Anterior Lumbar Plate: Fixed Screws vs. Variable Screws
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to slow enrollment
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-016
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Degenerative Disc Disease; Spinal Stenosis; Spondylolisthesis
Keywords: Degenerative Disc Disease; Spinal Stenosis; Spondylolisthesis; ALIF; fusion success; Anterior Lumbar Plate; fixed versus variable screw configurations; Anterior Lumbar Interbody Fusion to treat spinal instability
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spinal Stenosis; Spondylolisthesis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Trinica Anterior Lumbar Plate System with fixed screws only
  Interventions: Device: Trinica Anterior Lumbar Plate System
- Group 2 (Experimental): Trinica Anterior Lumbar Plate System with variable screws only
  Interventions: Device: Trinica Anterior Lumbar Plate System
- Group 3 (Experimental): Trinica Anterior Lumbar Plate with hybrid screw configuration (2 fixed-angle screws with 2 variable-angle screws).
  Interventions: Device: Trinica Anterior Lumbar Plate System

INTERVENTIONS:
Device: Trinica Anterior Lumbar Plate System — Trinica Anterior Lumbar Plate System accommodates the use of either fixed- or variable-angle screws. This study is a comparison of clinical outcomes from anterior lumbar interbody fusion patients receiving the Trinica Anterior Lumbar Plate system with either all fixed-angle screws, variable-angle screws, or a hybrid configuration.

SUMMARY:
Trinica Anterior Lumbar Plate (ALP) System is a commercially available, supplemental fusion device for use in the lumbar or sacral spine (L1-S1) to treat instability. The system provides the surgeon with the ability to supplement an interbody device with anterior plate fixation. The device's bone-plate interface is enhanced through use of fixed-angled screws,variable-angle screws or a combination of both to accommodate various combinations of screw configurations, resulting in enhanced fixation tailored to individual patient needs. Clinical outcomes data, including a comparison of different screw configurations, is needed to support the use and of the Trinica ALP System.

DETAILED DESCRIPTION:
In the cervical spine, literature shows that a static plate utilizing fixed screws loses its ability to load share and to limit motion following subsidence of the interbody spacer. In contrast, a dynamic plate system utilizing variable-angle screws maintains load-sharing and stiffness following subsidences. Increasing the load on the bone graft in the interbody space increases the rate of graft fusion. Although literature exists supporting the in vivo use of anterior cervical plate systems and the advantages of screw angulation, there is no data evaluating and supporting the use of anterior plate systems in the lumbar spine. The different biomechanical loads between cervical and lumbar spine suggest cervical data may not generalize to the lumbar spine. Additionally, it will be useful to characterize the effect of different screw configurations on subsidence and stress shielding and fusion success. The proposed study will not only assess clinical outcomes following Trinica ALP implantation, but will also provide valuable comparison data regarding two different screw configurations.

The study is a prospective, randomized, between groups design. The subject pool will be comprised of individuals who are appropriate for spinal fusion surgery, and who meet the inclusion criteria. Subjects will be randomly assigned to one of three screw configurations. All subjects will receive structural allograft (Puros A Anterior Allograft) as interbody support. Other procedures identified by the surgeon to be in the best interest of the patient may be completed but are not required by the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Spinal stenosis
* Spondylolisthesis Degenerative disc disease (defined as back pain of discogenic origin with degeneration of the disc confirmed by history and radiographic studies)
* Fracture (including dislocation or subluxation)
* Spine tumor
* Scoliosis
* Lordotic deformities of the spine

Exclusion Criteria:

* An active systemic or local infection
* Previous fusion attempt at index level
* A local inflammation with or without fever or leukocytosis
* Pregnancy
* Obesity (BMI >40 kg/m2)
* Drug or alcohol abuse
* Uncooperativeness or neurological or mental illness rendering the individual unwilling or unable to follow instructions
* Inability to restrict high activity level
* A suspected or documented metal allergy or intolerance
* A poor prognosis for good wound healing (e.g., decubitus ulcer, end-stage diabetes, severe protein deficiency and/or malnutrition)
* Any medical or surgical condition that would preclude the potential benefit of spinal implant surgery, prevent secure component fixation, or seriously increase the risk of tolerating any surgical procedure,
* Any other "contraindications" as enumerated in the device's "Instructions for Use".

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Alabama Spine Institute, Daphne, Alabama
  - Ronderos Neurosurgery Center, Mobile, Alabama
  - Loma Linda University Orthopedic Center, San Bernardino, California

RESULTS

PARTICIPANT FLOW:
Groups:
- ALP With Fixed Screws: Trinica Anterior Lumbar Plate System with fixed screws only
  Trinica Anterior Lumbar Plate System: Trinica Anterior Lumbar Plate System accommodates the use of either fixed- or variable-angle screws. This study is a comparison of clinical outcomes from anterior lumbar interbody fusion patients receiving the Trinica Anterior Lumbar Plate system with either all fixed-angle screws, variable-angle screws, or a hybrid configuration.
- ALP With Variable Screws: Trinica Anterior Lumbar Plate System with variable screws only
  Trinica Anterior Lumbar Plate System: Trinica Anterior Lumbar Plate System accommodates the use of either fixed- or variable-angle screws. This study is a comparison of clinical outcomes from anterior lumbar interbody fusion patients receiving the Trinica Anterior Lumbar Plate system with either all fixed-angle screws, variable-angle screws, or a hybrid configuration.
- ALP With Hybrid Screws: Trinica Anterior Lumbar Plate with hybrid screw configuration (2 fixed-angle screws with 2 variable-angle screws).
  Trinica Anterior Lumbar Plate System: Trinica Anterior Lumbar Plate System accommodates the use of either fixed- or variable-angle screws. This study is a comparison of clinical outcomes from anterior lumbar interbody fusion patients receiving the Trinica Anterior Lumbar Plate system with either all fixed-angle screws, variable-angle screws, or a hybrid configuration.
Period: Overall Study
Arm/Group | ALP With Fixed Screws | ALP With Variable Screws | ALP With Hybrid Screws
Started | 5 | 11 | 3
Completed | 0 | 6 | 0
Not Completed | 5 | 5 | 3
Not completed — Study Terminated slow enrollement | 5 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 5 | 11 | 3 | 19
Age, Continuous [Mean (Full Range); unit: Years] | 54 [45 to 66] | 51 [35 to 74] | 45 [33 to 55] | 51 [33 to 74]
Sex: Female, Male [Count of Participants; unit: Participants] — Number
  Participants
    Female | 1 | 6 | 1 | 8
    Male | 4 | 5 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: Clinical Outcomes (Oswestry Disability Index, SF-12, Numeric Pain Rating Scale, Surgeon Assessment, Patient Self Assessment, Radiological Assessment)
Description: - Fusion Assessment
Time Frame: Pre-operative, Operative; Follow-ups at 3 Months, 6 Months, 12 Months, and 24 Months
Population: Data not analyzed because study was stopped due to slow enrollment.
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2 | Group 3
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/11 | 0/3
Other Adverse Events (participants affected / at risk) | 4/5 | 4/11 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=5) | Group 2 (N=11) | Group 3 (N=3)
Cervical Disc Disease (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 — Pt. developed cervical disc disease, had surgery for cervical fusion
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=5) | Group 2 (N=11) | Group 3 (N=3)
Illeus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (General disorders) | 2 (2) | 1 (1) | 0 (0)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — Incision site infection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No